CLINICAL TRIAL: NCT02126501
Title: Randomized Control Trial of Weaning NCPAP From Preterm Infants: Sudden Wean Versus Weaning by Gradually Decreasing Pressure
Brief Title: Comparing Weaning of Nasal Continuous Positive Airway Pressure (CPAP) From Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC 13/01/VA03
Record Dates: First submitted 2014-03-17; First posted 2014-04-30 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Respiratory Distress Syndrome
Keywords: weaning; NCPAP; Preterm; sudden wean; gradual pressure off wean
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sudden wean (No Intervention): When ready Nasal Continuous Positive Airway Pressure (NCPAP) will be removed from the neonate
- Gradual pressure wean (Active Comparator): NCPAP will be removed by gradually decreasing pressure over 24 hours once the weaning is decided
  Interventions: Other: Gradual pressure wean

INTERVENTIONS:
Other: Gradual pressure wean — NCPAP will be removed by gradually decreasing pressure over 24 hours once the weaning is decided
  Arms: Gradual pressure wean

SUMMARY:
To compare the 2 methods of weaning of nasal continuous positive airway pressure (CPAP) in premature babies born between 26 and 32 weeks

DETAILED DESCRIPTION:
To study the weight and the post menstrual age (PMA) at the time of NCPAP wean utilizing the method of sudden wean as compared to gradual wean.

Methods: A prospective randomized trial was conducted comparing sudden weaning with gradual weaning from NCPAP in neonates with gestational age between 26 and 32 weeks. The patients were randomized to one of the two methods of weaning from NCPAP and their success was compared

ELIGIBILITY:
Inclusion Criteria:

* All neonates born 26 to 32 weeks of gestational age

Exclusion Criteria:

* Those with severe congenital anomalies and chromosomal defects including congenital heart disease, neurological malformations, chest and airway abnormalities and lung hypoplasia

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Success of weaning on first trial off NCPAP | Completion of Nasal Continuous Positive Airway Pressure (NCPAP) treatment, expected average of 4 weeks

SECONDARY OUTCOMES:
Weight and corrected GA when come off oxygen | when off supplemental oxygen expected average of 2 weeks
Weight and corrected gestational age (GA) when neonates could come off NCPAP | Completion of Nasal Continuous Positive Airway Pressure (NCPAP) treatment, expected average of 4 weeks

OTHER OUTCOMES:
length of stay in the neonatal intensive care unit | when ready to be discharged, expected average of 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu Rastogi, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides medcial center, Brooklyn, New York, United States

REFERENCES:
- [Derived] Amatya S, Macomber M, Bhutada A, Rastogi D, Rastogi S. Sudden versus gradual pressure wean from Nasal CPAP in preterm infants: a randomized controlled trial. J Perinatol. 2017 Jun;37(6):662-667. doi: 10.1038/jp.2017.10. Epub 2017 Feb 23. PMID 28230835